CLINICAL TRIAL: NCT02017847
Title: Assessment of Intensity Cut Off Points for Physical Activity Measured by Activity Monitors in Elderly Persons
Brief Title: Intensity of Physical Activity Measured by Activity Monitors in Elderly Persons
Acronym: GEN100
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: GEN100Study5
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Healthy
Keywords: oxygen consumption; activity monitors; METs; intensity

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Gen100: 150 participants in the Generation 100 study with anticipated 3000 participants aged 70-75

SUMMARY:
Aim of this study is to identify intensity cut off points for physical activity in a population over the age of 70.

DETAILED DESCRIPTION:
Activity monitors measure activity in counts. The higher the counts, the higher the intensity of the measured activity. In this study the count cut off points for low, moderate and high intensity activity will be investigated in a population of elderly people over the age of 70. This information will subsequently (in future studies) be used to investigate the physical activity patterns in a population of elderly over the age of 70 who have worn an activity monitor for a duration of 7 days.

ELIGIBILITY:
Inclusion Criteria:

* ability to walk at least 1km,
* born in 1938,1939,1940,1941 or 1942
* Sufficiently good health to be able to take part in the study, as determined by the researchers

Exclusion Criteria:

* Illness or disability that precludes exercise or hinders completion of the study
* Uncontrolled hypertension
* Symptomatic valve disease
* hyper tropic cardio-myopathy
* unstable angina
* Active cancer
* Test results indicating that study participation is unsafe
* Inclusion in other studies conflicting with participation in this one

Ages: 70 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Persons in the age of 70-76 living in Trondheim, Norway
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2013-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Intensity of physical activity | 1 year
  measured in counts by activity monitors

CONTACTS AND LOCATIONS:
Overall Officials: Nina Zisko, MSc, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- NTNU, Faculty of Medicine Department, of Circulation and Medical Imaging, Trondheim, Norway

REFERENCES:
- [Result] Zisko N, Carlsen T, Salvesen O, Aspvik NP, Ingebrigtsen JE, Wisloff U, Stensvold D. New relative intensity ambulatory accelerometer thresholds for elderly men and women: the Generation 100 study. BMC Geriatr. 2015 Aug 4;15:97. doi: 10.1186/s12877-015-0093-1. PMID 26238198
- See also: Generation 100 — http://www.ntnu.edu/cerg/generation100